CLINICAL TRIAL: NCT03443375
Title: Effects of Resistance Training Periodization on Hemodynamic, Morphofunctional and Cognitive Parameters of Robust Older Women.
Brief Title: Exercise Periodization and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Hélio José Coelho Júnior, Mr. Coelho-Junior, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 835.733
Record Dates: First submitted 2018-02-08; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Aging; Physical Activity; Sarcopenia; Cognitive Decline; Blood Pressure; Physical Disability
Keywords: Older adults; Physical function; Muscle mass; Short-term memory; Executive function; Blood Pressure; Resistance training; Exercise training; Periodization
MeSH Terms: conditions — Motor Activity; Sarcopenia; Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nonperiodized resistance training (Experimental): The Nonperiodized group performed was an intervention based on resistance exercise program with a constant intensity.
  Interventions: Other: Physical exercise
- Daily undulating periodized (Experimental): The Daily undulating periodized program was an intervention based on daily alterations on exercise load. .
  Interventions: Other: Physical exercise
- Control group (No Intervention): The control group remained their regular habits of life during all study period, without engaging in physical exercise programs.

INTERVENTIONS:
Other: Physical exercise — The interventions proposed in the present trial were based on a safe and well-established exercise training program
  Arms: Daily undulating periodized; Nonperiodized resistance training

SUMMARY:
The present study aimed at investigating the effects of two different resistance training protocols - nonperiodized (NP) and daily undulating periodization (DUP) - on hemodynamic, morphofunctional and cognitive parameters of robust older women. Methods: Forty-two older women were randomized allocated into one of the three experimental groups: NP, DUP, and control group (CG). Evaluations of the hemodynamic, morphofunctional and cognitive parameters occurred before, during and after six months. The exercise groups performed the program of exercise twice a week over 22 weeks. In NP, the two weekly sessions were based on 3 sets of 8-10 repetitions at a difficult intensity. However, in DUP, a power exercise session based on 3 sets of 8-10 repetitions at a moderate intensity was added in the first session of the week.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥60 years;
* Female;
* Not having been part of a systematic program of physical exercises in the last 6 months;
* MEEM score >19 points;
* Kihon checklist score >10 points;
* Capacity to perform the basic and instrumental activities of daily living according to Katz and Pfeffer indexes;
* Self-reported good memory;
* Complete all measurements.

Exclusion Criteria:

* Changes on antihypertensive medication in the past 6 months prior to inclusion in the study;
* Cardiovascular disease (i.e., acute myocardial infarction, stroke, peripheral arterial disease, and transient ischemic disease)
* Metabolic disease (i.e., diabetes mellitus type I or II), pulmonary disease (i.e., emphysema)
* Neurological and/or psychiatric disease (i.e., Parkinson's or Alzheimer's disease)
* Skeletal muscle disorders
* Comorbidities associated with greater risk of falls
* Recent history of smoking or alcohol abuse
* Hormone replacement therapy and/or psychotropic drugs.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in transfer capacity in seconds | 6 months
  TUG performance

SECONDARY OUTCOMES:
Changes in fat-free mass in kg | 6 months
  Fat-free mass
Changes in overall cognitive capacity in points | 6 months
  MEEM
Changes in blood pressure in mmHg | 6 months
  Blood Pressure
Changes in shor-term memory in points | 6 months
  Memory

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coelho-Junior HJ, Goncalves IO, Camara NOS, Cenedeze MA, Bacurau RF, Asano RY, Santana J, Caperuto E, Uchida MC, Rodrigues B. Non-periodized and Daily Undulating Periodized Resistance Training on Blood Pressure of Older Women. Front Physiol. 2018 Nov 27;9:1525. doi: 10.3389/fphys.2018.01525. eCollection 2018. PMID 30542289